CLINICAL TRIAL: NCT01042041
Title: A Phase 1 Study of Sorafenib Integrated With Chemoembolization for Patients With Unresectable Hepatocellular Carcinoma
Brief Title: Sorafenib Tosylate and Chemoembolization in Treating Patients With Unresectable Liver Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Soulen, Michael, Abramson Cancer Center of The University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 08208; NCI-2009-01488
Record Dates: First submitted 2009-12-10; First posted 2010-01-05 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer; Localized Unresectable Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Sorafenib; Doxorubicin; Cisplatin; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive oral sorafenib tosylate twice daily. Beginning 2 weeks later, patients undergo chemoembolization with cisplatin, doxorubicin hydrochloride, and mitomycin C. Chemoembolization repeats once a month for up to 4 procedures in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sorafenib tosylate; Drug: doxorubicin hydrochloride; Drug: cisplatin; Drug: mitomycin C; Procedure: transarterial chemoembolization; Procedure: hepatic artery embolization

INTERVENTIONS:
Drug: sorafenib tosylate — Given orally
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Drug: doxorubicin hydrochloride — Given via transarterial/hepatic chemoembolization
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF; Adriblastina
Drug: cisplatin — Given via transarterial/hepatic chemoembolization
  Other Names: CACP; CDDP; CPDD; DDP; Neoplatin; PDD
Drug: mitomycin C — Given via transarterial/hepatic chemoembolization
  Other Names: MITC; MITO; MITO-C; Mito-Medac; Mitocin-C; MTC
Procedure: transarterial chemoembolization
  Other Names: TACE
Procedure: hepatic artery embolization

SUMMARY:
RATIONALE: Sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth or by blocking blood flow to the tumor. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Chemoembolization kills tumor cells by blocking the blood flow to the tumor and keeping chemotherapy drugs near the tumor.

PURPOSE: This phase I trial is studying side effects and best dose of sorafenib tosylate when given together with chemoembolization in treating patients with unresectable liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the toxicity and safety of integrating sorafenib with chemoembolization for unresectable hepatocellular carcinoma.

SECONDARY OBJECTIVE:

I. To observe the imaging response (AASLD/EASL modification of RECIST) and time to progression following chemoembolization in conjunction with sorafenib.

OUTLINE:

Patients receive oral sorafenib tosylate twice daily. Beginning 2 weeks later, patients undergo chemoembolization with cisplatin, doxorubicin hydrochloride, and mitomycin C.

Chemoembolizaton repeats once a month for up to 4 procedures in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 4 weeks and then every 3 months.

ELIGIBILITY:
Inclusion

* Histologically confirmed hepatocellular carcinoma
* AND/OR Magnetic Resonance Imaging (MRI) or Computerized Tomography (CT) consistent with liver cirrhosis AND at least one solid liver lesion > 2cm with arterial-phase enhancement and delayed washout regardless of alpha-feto protein levels (AFP)
* AND/OR AFP > 400ng/mL AND evidence of at least one solid liver lesion > 2cm regardless of specific imaging characteristics on CT or MRI
* Patient is not a candidate for transplantation, resection, or ablation; for whom the intended therapy is chemoembolization
* Patient meets clinical criteria for treatment with chemoembolization
* Absolute contraindications to chemoembolization include an uncorrectable bleeding disorder, uncorrectable contrast sensitivity, leukopenia (white blood cell count < 1000/uL), cardiac or renal insufficiency (serum creatinine > 2.0mg/dL), hepatic encephalopathy, jaundice, or dilated intrahepatic bile ducts
* Portal vein occlusion is a relative contraindication and chemoembolization can be performed only if there are collateral vessels with hepato-pedal flow demonstrated angiographically
* Hepatic compromise as determined by the following combination of parameters is a contraindication to therapy: lactate dehydrogenase > 425 U/L, aspartate aminotransferase > 100 U/L, total bilirubin > 2.0 mg/dL and > 50% liver volume replaced by tumor
* Patients may have been treated with ablation or resection in the past, but no sooner than 4 weeks before study registration
* Patients may NOT have been previously treated with sorafenib, chemoembolization, radioembolization, or systemic chemotherapy with cytotoxic agents or molecularly targeted agents
* ECOG performance status =< 2
* Life expectancy of greater than 3 months
* Platelets >= 50,000/mcL
* Total bilirubin =< 2.0 mg/dl
* AST(SGOT)/ALT(SGPT) =< 3X institutional upper limit of normal
* Creatinine =< 1.5 mg/dl
* INR =< 1.5
* Patients must have no clinical signs of heart failure and meet New York Heart Association functional classification I or II defined as:

Class I - Patients with no limitation of activities; they suffer no symptoms from ordinary activities; Class II - Patients with slight, mild limitation of activity; they are comfortable with rest or with mild exertion

* Because agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion

* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sorafenib
* History of radiologic contrast reactions not controlled by standard premedications
* Patients must not be taking cytochrome P450 enzyme inducing drugs
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study
* Breastfeeding should be discontinued
* Prophylactic use of G-CSF or GM-CSF is not permitted on this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Dose adjustment, number and percentage of subjects with adverse events, laboratory changes, number and percentage of subjects with laboratory values that are outside the pre-determined ranges, cumulative toxicity, and TLT. | 8 months

SECONDARY OUTCOMES:
Time to Disease Progression | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Soulen, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania, United States